CLINICAL TRIAL: NCT01102335
Title: The Observation Of Safety And Survival Of Hepatocellular Carcinoma After Transcatheter Arterial Chemoembolization Combined With Anti-hepatitis B Virus Therapy
Brief Title: Synergistic Treatment for Hepatocellular Carcinoma (HCC) Using Transcatheter Arterial Chemoembolization (TACE) With Anti-hepatitis B Virus (Anti-HBV) Therapy
Acronym: TACEHBV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Professor Jing-lin Xia, Liver Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI-001
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatitis B virus; Antiviral Agents; Liver Neoplasms; Drug Toxicity; Survival
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Liver Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telbivudine (Experimental)
  Interventions: Procedure: Transcatheter arterial chemoembolization (TACE); Drug: Telbivudine
- TACE only (Active Comparator)
  Interventions: Procedure: Transcatheter arterial chemoembolization (TACE)

INTERVENTIONS:
Procedure: Transcatheter arterial chemoembolization (TACE) — The procedure is performed under local anaesthesia. The femoral artery at groin region is punctured for arterial access. Angiography is performed for demonstration of vascular structures before embolization.The arteries supplying the tumor are selectively catheterized, this includes the hepatic arteries or other extrahepatic collateral arteries.The chemotherapeutic agent(s) is mixed with lipiodol (an oily contrast) to enhance tumour uptake. Following delivery of the lipiodol/chemotherapy mixture, small gelfoam particles may be injected to reinforce the effect of treatment.
Drug: Telbivudine — anti-HBV drug
  Other Names: Sebivo
  Arms: Telbivudine

SUMMARY:
The purpose of this study is to elucidate the influence of anti-hepatitis B virus therapy on safety and survival of HCC patient after transcatheter arterial chemoembolization.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma
* treated with transcatheter arterial chemoembolization (TACE)
* HBVDNA > 10^3copies/mL, including alanine aminotransferase (ALT) normal patient
* expected survive time > 1 year
* HBV marker positive (anyone of HbsAg, HbsAb, HbeAg, HbeAb and HbcAb)

Exclusion Criteria:

* antiviral therapy history
* alanine aminotransferase (ALT) >400 U/L
* serum total bilirubin > 50 μmol/L
* HBVDNA > 10^9copies/mL
* extrahepatic metastasis or main portal vein embolus
* apparent cardiac or pulmonary dysfunction
* liver function: Child B or Child C
* HCV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months

SECONDARY OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: jinglin xia, MD, Principal Investigator — Liver cancer institute, Zhongshan Hospital
Locations (1):
- Liver cancer institute, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China